CLINICAL TRIAL: NCT03916341
Title: Smoking and Ventricular Repolarization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Tobacco Related Disease Research Program (Other)
Responsible Party: Principal Investigator, Holly R Middlekauff, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 19-000452
Record Dates: First submitted 2019-04-10; First posted 2019-04-16 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Sudden Cardiac Death; Prolonged QTc Interval
Keywords: e-cigarettes; tobacco cigarettes; nicotine; ventricular repolarization
MeSH Terms: conditions — Death, Sudden, Cardiac; Vaping | interventions — Nicotine

STUDY DESIGN:
Intervention Model Description: Crossover with 4 week washout
Who Masked: Outcomes Assessor
Masking Description: Single (outcomes assessor) code
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-user (Experimental): Non- users will use, in a randomized, crossover fashion with a 4 week washout, an 1) EC with nicotine, 2) EC without nicotine, and 3) an empty EC (control)
  Interventions: Other: EC with nicotine; Other: EC without nicotine; Other: control
- Chronic EC user (Experimental): Chronic EC users will use, in a randomized, crossover fashion with a 4 week washout, an 1) EC with nicotine, 2) EC without nicotine, and 3) an empty EC (control)
  Interventions: Other: EC with nicotine; Other: EC without nicotine; Other: control
- Chronic TC smoker (Experimental): Chronic TC smokers will use, in a randomized, crossover fashion with a 4 week washout, a 1) TC with nicotine (own brand), 2) research TC with very low level nicotine, and 3) a straw (control)
  Interventions: Other: control; Other: TC with nicotine (own brand); Other: research TC with very low level nicotine

INTERVENTIONS:
Other: EC with nicotine — Use an EC with nicotine for up to 30 minutes
  Arms: Chronic EC user; Non-user
Other: EC without nicotine — Use an EC without nicotine for up to 30 minutes
  Arms: Chronic EC user; Non-user
Other: control — sham control
Other: TC with nicotine (own brand) — smoke a TC
  Arms: Chronic TC smoker
Other: research TC with very low level nicotine — smoke a research TC with very low level nicotine
  Arms: Chronic TC smoker

SUMMARY:
Randomized controlled trial of acute use of electronic cigarette or tobacco cigarette on parameters of ventricular repolarization.

DETAILED DESCRIPTION:
Non-user or chronic electronic cigarette (EC) users will use an EC or control on three occasions:1) EC with nicotine, 2) EC without nicotine, 3) empty EC (control).

Chronic tobacco cigarette (TC) smokers will use a TC or control on three occasions: 1) TC with nicotine (subject's own brand), 2) research TC with very low nicotine, 3) straw (control). The electrocardiogram will be recorded before and after acute exposures and analyzed for parameters representative of ventricular repolarization.

ELIGIBILITY:
Inclusion Criteria:

* Healthy non-smokers chronic TC smokers (non-e-cig users) Chronic EC smokers (Non-TC smokers)

Exclusion Criteria:

* Cardiac disease, respiratory disease, diabetes

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Tpe | Change in Tpe 5 minutes before and 5 minutes after cigarette use
  interval indicative of ventricular repolarization measured on ECG
Tpe/QT | Change in Tpe/QT 5 minutes before and 5 minutes after cigarette use
  ratio of intervals indicative of ventricular repolarization measured on ECG
Tpe/QTc | Change in Tpe/QTc 5 minutes before and 5 minutes after cigarette use
  ratio of intervals indicative of ventricular repolarization measured on ECG

SECONDARY OUTCOMES:
QT | Change in QT 5 minutes before and 5 minutes after cigarette use
  interval indicative of ventricular repolarization measured on ECG
QTc | Change in QTc 5 minutes before and 5 minutes after cigarette use
  interval indicative of ventricular repolarization measured on ECG

CONTACTS AND LOCATIONS:
Locations (1):
- UCaliforniaLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No